CLINICAL TRIAL: NCT01484275
Title: A Phase 2, Randomized, Blinded, Placebo-controlled, Multicenter Study of Siltuximab (Anti IL 6 Monoclonal Antibody) in Subjects With High-risk Smoldering Multiple Myeloma
Brief Title: A Study of Siltuximab (Anti- IL 6 Monoclonal Antibody) in Patients With High-risk Smoldering Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100755; CNTO328SMM2001 (Other: Janssen Research & Development, LLC); 2011-001735-22 (EudraCT Number); NCT01563666 (obsolete NCT alias)
Record Dates: First submitted 2011-12-01; First posted 2011-12-02 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: High-risk Smoldering Multiple Myeloma
Keywords: High-risk smoldering multiple myeloma; Multiple myeloma; Siltuximab
MeSH Terms: conditions — Multiple Myeloma | interventions — siltuximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Siltuximab (Experimental): Type=exact, unit=mg/kg, number=15, form=intravenous infusion, route=intravenous use, every 4 weeks until progression to symptomatic multiple myeloma, unacceptable toxicity, withdrawal of consent, or the end of the study.
  Interventions: Drug: Siltuximab
- Placebo (Placebo Comparator): Form=intravenous infusion, route=intravenous use route=intravenous, use every 4 weeks until progression to symptomatic multiple myeloma, unacceptable toxicity, withdrawal of consent, or the end of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Siltuximab — Type=exact, unit=mg/kg, number=15, form=intravenous infusion, route=intravenous use, every 4 weeks until progression to symptomatic multiple myeloma, unacceptable toxicity, withdrawal of consent, or the end of the study.
  Arms: Siltuximab
Drug: Placebo — Form=intravenous infusion, route=intravenous use route=intravenous, use every 4 weeks until progression to symptomatic multiple myeloma, unacceptable toxicity, withdrawal of consent, or the end of the study.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of siltuximab compared with placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial) in patients with high-risk smoldering multiple myeloma (SMM).

DETAILED DESCRIPTION:
This is a randomized (treatment assigned by chance), double-blind (neither patient nor investigator know which treatment is given), multicenter study to evaluate the safety and efficacy of siltuximab compared with placebo in patients with high-risk SMM (defined as bone marrow plasma cells >=10% and either serum monoclonal protein >=3 g/dL, or abnormal free light chain ratio <0.126 or >8 and serum M-protein <3 g/dL but >=1 g/dL). Approximately 74 patients will receive either siltuximab or placebo by intravenous (IV, injection into a vein) infusion every 4 weeks until progression to symptomatic multiple myeloma, unacceptable toxicity, withdrawal of consent, or the end of the study (approximately 4 years after randomization of the last patient). Efficacy, pharmacokinetics, immunogenicity, and potential biomarkers will be assessed at time points defined in the protocol. Patient reported outcomes (European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire-Core 30, Brief Pain Inventory [worst pain], Non-Chemotherapy Anemia Symptom Scale) will be administered before any procedure or treatment at each visit. Patient safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of smoldering multiple myeloma (SMM) for <4 years
* Diagnosis of high-risk SMM (defined as bone marrow plasma cells >=10% and either serum monoclonal protein >=3 g/dL, or abnormal free light chain ratio <0.126 or >8 and serum M-protein <3 g/dL but >=1 g/dL)
* Patients must be within certain limits for protocol-specified laboratory tests
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Women not of childbearing potential must be postmenopausal, permanently sterilized, or otherwise incapable of pregnancy
* Women of childbearing potential must agree to use adequate birth control measures and agree to not donate eggs for the purpose of assisted reproduction during the study and for 3 months after receiving the last dose of study agent, and must have a negative pregnancy test at screening
* Men must agree to use a double-barrier method of birth control and to not donate sperm during the study and for 3 months after receiving the last dose of study agent

Exclusion Criteria:

* Having symptomatic multiple myeloma, defined by any of the following (if due to myeloma): lytic bone lesions, severe osteopenia (low bone density), pathologic fractures, hypercalcemia (too much calcium in the blood), kidney insufficiency; symptomatic hyperviscosity of the blood, or recurrent serious bacterial infections such as pneumonia
* Primary systemic amyloid light (AL) chain amyloidosis (a build-up of amyloid light chain proteins in the blood)
* Prior or concurrent exposure to approved or investigational multiple myeloma treatments (concurrent treatment with bone-protecting agents (eg, bisphosphonates, denosumab), or steroids (not exceeding 10 mg prednisone per day or equivalent) are only allowed if given in a stable dose and for a nonmalignant condition; concurrent treatment with erythropoietin-stimulating agents (ESAs) are not allowed.)
* Prior exposure to agents targeting interleukin 6 (IL 6) or the IL 6 receptor
* Other malignancy within the past 3 years, except for the following, if treated and not active: basal cell or nonmetastatic (non-spreading) squamous cell carcinoma of the skin, cervical carcinoma or International Federation of Gynecology and Obstetrics Stage 1 carcinoma of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2015-05-12 (Actual); Study Completion 2019-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (40):
- United States (8):
  - Chicago, Illinois
  - Rockville, Maryland
  - Detroit, Michigan
  - New York, New York
  - Kittanning, Pennsylvania
  - Philadelphia, Pennsylvania
  - Greenville, South Carolina
  - Dallas, Texas
- Australia (3):
  - Camperdown
  - East Melbourne
  - Randwick
- Belgium (3):
  - Antwerp
  - Brussels
  - Ghent
- France (4):
  - Dijon
  - Nantes
  - Tours
  - Villejuif
- Germany (3):
  - Berlin
  - Hamburg
  - Heidelberg
- Athens, Greece
- Israel (6):
  - Ashkelon
  - Jerusalem
  - Nahariya
  - Netanya
  - Petah Tikva
  - Tel Aviv
- South Korea (2):
  - Daejeon
  - Seoul
- Spain (5):
  - Barcelona
  - Barcleona
  - Madrid
  - Salamanca
  - Valencia
- Sweden (3):
  - Gothenburg
  - Linköping
  - Stockholm
- United Kingdom (2):
  - London
  - Manchester

REFERENCES:
- [Derived] Brighton TA, Khot A, Harrison SJ, Ghez D, Weiss BM, Kirsch A, Magen H, Gironella M, Oriol A, Streetly M, Kranenburg B, Qin X, Bandekar R, Hu P, Guilfoyle M, Qi M, Nemat S, Goldschmidt H. Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of Siltuximab in High-Risk Smoldering Multiple Myeloma. Clin Cancer Res. 2019 Jul 1;25(13):3772-3775. doi: 10.1158/1078-0432.CCR-18-3470. Epub 2019 Mar 19. PMID 30890552

RESULTS

PARTICIPANT FLOW:
Groups:
- Siltuximab: Participants received 15 milligram per kilogram (mg/kg) of siltuximab as a 1-hour intravenous (IV) infusion every 4 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or the end of the study (up to 4 years after randomization of the last participant).
- Placebo: Participants received placebo as a 1-hour IV infusion every 4 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or the end of the study (up to 4 years after randomization of the last participant).
Period: Overall Study
Arm/Group | Siltuximab | Placebo
Started | 43 | 42
Completed | 0 | 0
Not Completed | 43 | 42
Not completed — Study terminated by sponsor | 28 | 32
Not completed — Other | 10 | 0
Not completed — Death | 3 | 4
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Siltuximab | Placebo | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (10.95) | 59.5 (12.03) | 61.4 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 26 | 22 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 35 | 37 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 4 | 4 | 8
  Belgium | 1 | 1 | 2
  France | 5 | 1 | 6
  Germany | 5 | 14 | 19
  Israel | 7 | 3 | 10
  Korea, Republic Of | 3 | 2 | 5
  Spain | 9 | 6 | 15
  United Kingdom | 4 | 2 | 6
  United States | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: One-Year Progression-Free Survival (PFS) Rate
Description: One-year PFS rate is defined as the percentage (%) of participants surviving 1 year after randomization without progression to multiple myeloma or death estimated by the Kaplan-Meier method and based on the International Myeloma Working Group (IMWG) calcium, renal, anemia, and bone lesions (CRAB) criteria. Progressive disease (PD) is defined as presence of an M- component in serum plus clonal plasma cells in the bone marrow plus 1 or more of the following: Calcium elevation (greater than [>] 11.5 milligram per deciliter [mg/dL] [> 2.88 millimoles per liter {mmol/L}]); Renal insufficiency (creatinine > 2 mg/dL [177 micromoles per liter or more]; Anemia (hemoglobin less than [<] 10 gram per deciliter [g/dL] or 2 g/dL lower than lower limit of normal [LLN] [hemoglobin < 6.5 mmol/L or 1.25 mmol/L lower than LLN]); Bone disease (lytic lesions or osteopenia).
Time Frame: Up to 1 Year
Population: Intent-to-treat (ITT) population included participants who were randomly assigned to siltuximab or placebo treatment group based on an integrated voice response system (IVRS).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 43 | 42
Percentage of participants | 84.5 [68.6 to 92.8] | 74.4 [57.3 to 85.5]

2. Secondary Outcome: Progressive Disease Indicator Rate (PDIR) at 6 Months
Description: PDIR is defined as percentage of participants who meet any of following criteria occurring within 6 months of start of treatment. a) CRAB criteria: true progression events, b) Serum M-protein: increase by 25 % compared with baseline at 2 consecutive assessments, c) Magnetic resonance imaging: unequivocal increase in focal bone lesions, d) Immunoparesis: decrease by 25% compared with baseline of 2 other non-affected immunoglobulin (Ig) (IgG, IgM, IgA) at 2 consecutive assessments, e) Hemoglobin: decrease of 1.5 g/dL (with at least 1 read below LLN) at 2 consecutive assessments, with no other identifiable cause. PD is defined as presence of M-component in serum plus clonal plasma cells in bone marrow plus 1 or more of following: Calcium elevation (> 11.5 mg/dL [> 2.88 mmol/L]); Renal insufficiency (creatinine >2 mg/dL [177 micro mol/L or more]); Anemia (hemoglobin <10 or 2 g/dL lower than LLN) [hemoglobin < 6.5 or 1.25 mmol/L lower than LLN]); Bone disease (lytic lesions or osteopenia).
Time Frame: At 6 Months
Population: Response evaluable population included participants who had a diagnosis of high-risk smoldering multiple myeloma (SMM) and received at least 1 dose of siltuximab/placebo treatment. In addition, participants were to have at least 1 post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 43 | 42
Percentage of participants | 30.2 [17.2 to 46.1] | 42.9 [27.7 to 59.0]

3. Secondary Outcome: Progression-Free Survival
Description: PFS is defined as the time between randomization and initial documented PD according to the CRAB - International Myeloma Working Group (IMWG) criteria or date of death, whichever occurs first. PD is defined as presence of an M-component in serum plus clonal plasma cells in the bone marrow plus 1 or more of the following: Calcium elevation (> 11.5 mg/dL [> 2.88 mmol/L]); Renal insufficiency (creatinine > 2 mg/dL [177 [micro mol/L or more]); Anemia (<10 g/dL or 2 g/dL) lower than LLN) [hemoglobin < 6.5 mmol/L or 1.25 mmol/L lower than LLN]); Bone disease (lytic lesions or osteopenia).
Time Frame: Up to 4.7 Years
Population: ITT population included participants who were randomly assigned to siltuximab or placebo treatment group based on an IVRS.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 43 | 42
Days | NA [703 to NA] — Here, NA signifies that median and upper limit of confidence interval (CI) was not estimable due to less number of events. | 715.0 [490 to 1232]

4. Secondary Outcome: Percentage of Participants With Serum M-protein Response
Description: Serum M-protein response is defined as a decrease of greater than or equal to (>=) 50% in serum M-protein compared with baseline at 2 consecutive assessments.
Time Frame: Up to 4.7 Years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 43 | 42
Percentage of participants | 2.3 [0.1 to 12.3] | 0.0 [0.0 to 8.4]

5. Secondary Outcome: Time to Worsening in European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire-Core 30 (EORTC-QLQ-C30) Scale Score
Description: Time to worsening in EORTC-QLQ-C30 (physical function scale) is defined as time between randomization and first documentation of a worsening in EORTC-QLQ-C-30. Worsening in the EORTC-QLQ-C30 is defined as 10 points decrease from baseline. It comprises module with 30 items. Questionnaire includes 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, nausea/vomiting), a global health and quality of life scale, and a number of single items assessing symptoms (dyspnea, loss of appetite, insomnia, constipation, diarrhoea). Instrument contains 28 items using a Likert scale with 4 response options: "Not at All," "A Little," "Quite a Bit," "Very Much" (scored 1-4). Two additional items use response options (1-7): 1=Very Poor, to 7=Excellent. All scale and item scores were linearly transformed to be in range from 0-100. A higher score represents a higher (better) level of functioning, or a higher (worse) level of symptoms.
Time Frame: Up to 4.7 Years
Population: ITT population included participants who were randomly assigned to siltuximab or placebo treatment group based on an IVRS who had 10 points decrease from baseline in the physical function scale.
Measure: Median (Full Range); unit: Days
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 22 | 21
Days | 125.50 [56.0 to 1021.0] | 118.00 [56.0 to 565.0]

6. Secondary Outcome: Time to Worsening in the Brief Pain Inventory (BPI) Worst Item Scores
Description: Time to worsening in the BPI worst item is defined as the time between randomization and the first documentation of a worsening in the BPI worst item. It has 2 domains reflecting pain severity and pain interference with domains of functioning and well-being. The selected item refers to the "worst" pain the patient has experienced over the past 24 hours. This item has been found to be most responsive to interference with key domains of functioning and well-being and may be used as a single item. Responses are provided on an 11-point numeric rating scale ranging from 0 "no pain" to 10 "pain as bad as you can imagine". Responses are described as mild (1 to 4), moderate (5 to 6) and severe (7 to 10). Worsening in the BPI worst item is defined as 2 points increase from baseline.
Time Frame: Up to 4.7 Years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 43 | 42
Days | 652.0 [226 to NA] — Here, NA signifies that upper limit of CI was not estimable due to an insufficient number of events. | 453.0 [277 to NA] — Here, NA signifies that upper limit of CI was not estimable due to an insufficient number of events.

7. Secondary Outcome: Number of Participants With Symptomatic Multiple Myeloma With Adverse Prognostic Features
Description: Number of participants who progressed to symptomatic multiple myeloma with stage III of International Staging System (ISS) or abnormal cytogenetic findings were assessed. The ISS system consists of stage I: beta2-microglobulin < 3.5 milligram per liter (mg/L) and albumin >= 3.5 gram (g)/100 ml; stage II: neither stage I nor stage III and stage III: beta2-microglobulin >= 5.5 mg/L.
Time Frame: Up to 4.7 Years
Population: The data was not collected and analyzed for this outcome measure as per the change in planned analysis.
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Best Response to First Subsequent Multiple Myeloma Treatment
Description: Best response to first subsequent anti-myeloma therapy was assessed by physician report at 6-month intervals and classified as: complete response (CR) (negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and < 5% plasms cells (PCs) in bone marrow); stringent CR (CR plus a normal FLC ratio, absence of clonal cells in bone marrow); near CR (< 5% PCs in a bone marrow aspirate, no increase in lytic bone lesions); very good partial response (VGPR) (serum and urine component detectable by immunofixation but not on electrophoresis, or >= 90% reduction in serum M-protein plus urine M-protein level <100 mg per 24 hour); partial response (PR): >= 50 reduction of serum M-protein, reduction in 24-hour urinary M-protein by >=90 % or to < 200 mg/24 hours); minimal response (>=25% but <= 49% reduction of serum M-protein and reduction in urine M-protein by 50%-89%); stable disease (not meeting criteria for CR, VGPR, PR, or PD); PD; not evaluable and unknown.
Time Frame: Up to 4.7 Years
Population: The data was not collected and analyzed for this outcome measure as per the change in planned analysis.
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time between randomization and death due to any cause.
Time Frame: Up to 4.7 Years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 43 | 42
Days | NA [NA to NA] — Here, NA signifies that median and confidence interval was not estimable due to less number of events. | NA [NA to NA] — Here, NA signifies that median and confidence interval was not estimable due to less number of events.

ADVERSE EVENTS:
Time Frame: Up to 4.7 Years
Description: Safety analysis set included participants who have received at least 1 administration of any study agent (siltuximab or placebo).
Arm/Group | Siltuximab | Placebo
All-Cause Mortality (participants affected / at risk) | 3/43 | 4/42
Serious Adverse Events (participants affected / at risk) | 13/43 | 13/42
Other Adverse Events (participants affected / at risk) | 41/43 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Siltuximab (N=43) | Placebo (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Eustachian Tube Disorder (Ear and labyrinth disorders) | 1 | 0
Gastric Disorder (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Pneumonia Streptococcal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Back Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Facial Paresis (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2
Oliguria (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 1
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Ischaemia (Vascular disorders) | 0 | 1
Poor Venous Access (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Siltuximab (N=43) | Placebo (N=42)
Anaemia (Blood and lymphatic system disorders) | 6 | 6
Neutropenia (Blood and lymphatic system disorders) | 8 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0
Palpitations (Cardiac disorders) | 1 | 4
Abdominal Distension (Gastrointestinal disorders) | 0 | 4
Abdominal Pain (Gastrointestinal disorders) | 3 | 6
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 5 | 7
Diarrhoea (Gastrointestinal disorders) | 6 | 7
Nausea (Gastrointestinal disorders) | 9 | 10
Stomatitis (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 8 | 3
Chest Pain (General disorders) | 1 | 5
Fatigue (General disorders) | 6 | 14
Influenza Like Illness (General disorders) | 1 | 5
Oedema Peripheral (General disorders) | 3 | 3
Pyrexia (General disorders) | 3 | 6
Bronchitis (Infections and infestations) | 3 | 3
Gastroenteritis (Infections and infestations) | 3 | 1
Herpes Zoster (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 9 | 15
Oral Herpes (Infections and infestations) | 0 | 4
Pneumonia (Infections and infestations) | 3 | 1
Rhinitis (Infections and infestations) | 1 | 4
Sinusitis (Infections and infestations) | 3 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 10
Urinary Tract Infection (Infections and infestations) | 3 | 3
Alanine Aminotransferase Increased (Investigations) | 4 | 0
Aspartate Aminotransferase Increased (Investigations) | 3 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 12
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 5
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 5 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 8
Dizziness (Nervous system disorders) | 3 | 6
Headache (Nervous system disorders) | 6 | 9
Sciatica (Nervous system disorders) | 4 | 2
Syncope (Nervous system disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 10
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 6 | 0
Hypertension (Vascular disorders) | 1 | 4

LIMITATIONS AND CAVEATS:
Siltuximab demonstrated positive trending toward 1-year PFS only in high risk SMM-group. Sponsor and Steering Committee decided not to further pursue clinical development of siltuximab for SMM and terminated study, and was considered as completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.